CLINICAL TRIAL: NCT04187482
Title: Functional and Cellular Benefits of Aerobic Exercise in Myotonic Dystrophy Type 1 Patients
Brief Title: Myotonic Dystrophy Type 1 Aerobic Exercise Study
Acronym: DM1ex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Mark Tarnopolsky, Principal Investigator, Professor, Director of Neuromuscular and Neurometabolic Clinic, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 7091
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Myotonic Dystrophy 1; Muscular Dystrophies
Keywords: aerobic exercise
MeSH Terms: conditions — Myotonic Dystrophy; Muscular Dystrophies | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants are undergoing 12-weeks of aerobic exercise training
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise training group (Experimental): All participants will be receiving same exercise training intervention
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — All participants with DM1 will undergo a 12-week aerobic exercise training intervention on a cycle ergometer

SUMMARY:
Myotonic dystrophy type 1 (DM1) is a genetic disease that primarily targets skeletal muscle resulting in severe weakness and muscle loss. As a result, individuals suffering from DM1 become very inactive and lose mobility resulting in a lower quality of life. This study will investigate the effect of a 12-week moderate intensity exercise protocol on skeletal muscle function and cellular benefits in DM1 patients.

DETAILED DESCRIPTION:
The present study is a repeated measures design, with sampling of the cohorts on two separate occasions. Upon obtaining informed consent, participants will be assigned into one of two groups:

Group 1: DM1 Exercise Group DM1 diagnosed, physically inactive males, n = 6 DM1 diagnosed, physically inactive females, n = 7

Group 2: Healthy controls (no exercise) Healthy, physically inactive males n = 6 Healthy, physically inactive females n = 7

Introduction - Day 1 (Visit 1); On the initial visit, the potential participant will come to McMaster Children's Hospital to meet with a study coordinator involved in the project. The coordinator will explain the study in detail, answer any questions, and review the consent form. Upon obtaining informed consent, eligible participants will complete a medical screening questionnaire to determine their readiness to perform exercise. Participant characteristics will then be measured. At this time, anthropometric measurements (i.e., height, weight, waist circumference) and a dual energy x-ray absorptiometry (DXA) measurement will be performed. This must be done in order to verify that the participant meets the inclusion criteria of being normal weight (BMI 18.5 - 24.9 kg/m2) or overweight (BMI 25 - 29.9 kg/m2). Following this screening, participants will undergo an ECG to measure any conductance blockage and perform a maximal cycling test to determine their aerobic capacity (V02max). Maximal aerobic testing will then be followed by another 12 lead ECG to detect any possible structural cardiac issues in our participants. Thereafter, participants will begin the following the study timeline, all of which will occur at the McMaster Children's Hospital, 2H Neurometabolic Clinic.

Baseline testing - Day 3 (Visit 2); Participants will arrive the following day to undergo functional testing which will include 6-minute walk test, 5x sit to stand, timed up and go, grip strength and maximal voluntary knee extension using the Biodex dynamometer. Participants will then complete the SF-36.

Follow up testing - Day 5 (Visit 3); Participants will arrive following an overnight fast (including no caffeine for 12 hours) and having abstained from any exercise for the prior 24 hours. Participants will undergo a muscle biopsy from the vastus lateralis.

DM1 participants only:

Exercise training - Visit 4 - 39; Participants will begin the exercise protocol consisting of 3 exercise sessions per week for a 12-week period. All exercise sessions will be done on a cycle ergometer (Lode, Groningen, Netherlands). Each exercise session will consist of 3 minutes of warm up, 30 minutes at 65% V02max and will end with 2 minutes of cool down. Exercise progression over the 12 weeks will go as follows:

* Weeks 1 and 2: 3 min warm up, 65% VO2max for 30 min, 2 min cool down
* Weeks 3 and 4: increase to 35 min (+ warm up/cool down)
* Weeks 5 and 6: drop to 30 min and increase to 70% VO2max
* Weeks 7 and 8: increase to 35 min (+ warm up/cool down)
* Weeks 9 and 10: drop to 30 min and increase to 75%VO2 max
* Weeks 11 and 12: increase to 35 min (+ warm up/cool down)

Endpoint testing - Visit 40; At this time, anthropometric re-measurements (i.e., height, weight, waist circumference) and a dual energy x-ray absorptiometry (DXA) measurement will be performed. Thereafter, participants will undergo an ECG to measure any conductance blockage and perform a maximal cycling test to determine their aerobic capacity (V02peak). Maximal aerobic testing will then be followed by another 12 lead ECG to detect any possible structural cardiac issues in our participants.

Endpoint testing - Visit 41; Participants will arrive the following day to undergo functional testing which will include 6-minute walk test, timed up and go, grip strength and maximal voluntary knee extension using the Biodex dynamometer. Participants will then complete the SF-36.

Endpoint testing - Visit 42; Participants will arrive following an overnight fast (including no caffeine for 12 hours) and having abstained from any exercise for the prior 24 hours. Participants will undergo a muscle biopsy from the vastus lateralis.

ELIGIBILITY:
Inclusion Criteria:

DM1 participants:

* Male or female clinically diagnosed with DM1
* CTG repeats 100-1000
* Normal weight (BMI 18.5 - 24.9 kg/m2) or overweight (BMI 25 - 29.9 kg/m2)

Age matched controls:

* Healthy men and women
* Normal weight (BMI 18.5 - 24.9 kg/m2) or overweight (BMI 25 - 29.9 kg/m2)
* Physically inactive (< 1-2 hour of formal exercise/week)

Exclusion Criteria:

* Smoking
* Obese (BMI > 30.0 kg/m2)
* Use of narcotic analgesic or anti-inflammatory drugs
* Type 1 or 2 diabetes (more than one anti-diabetic drug)
* Cardiovascular disease (recent myocardial infarction (< 6 months))
* Uncontrolled hypertension requiring more than 2 medications
* Congestive heart failure requiring more than one medication for control-
* Known liver disease
* Cognitive impairments limiting ability to provide informed consent
* Active musculoskeletal injuries and/or severe osteoarthritis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-03-29 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Maximal aerobic capacity | 3 months from enrolment
  VO2max in mL/min/kg-1

SECONDARY OUTCOMES:
6 minute walk test | 3 months from enrolment
  changes in number of meters walked during the 6 minute walk test
5x sit to stand | 3 months from enrolment
  changes in the time (seconds) needed to complete 5x sit to stand from a chair
timed up and go | 3 months from enrolment
  changes in the time (seconds) needed to complete a timed up and go test
Leg muscle strength | 3 months from enrolment
  maximal isometric knee extension via Biodex in N*m
Grip strength | 3 months from enrolment
  changes in grip strength (kg) using a hand dynamometer
Body composition | 3 months from enrolment
  change in fat free mass and fat mass measured via DXA in kg
Muscle fibre cross sectional area | 3 months after intervention is complete
  changes in fibre cross sectional area from muscle biopsy of vastus lateralis using immunoflourescence
Mitochondrial protein content | 3 months after intervention is complete
  changes in mitochondrial proteins from muscle biopsy of vastus lateralis using western blotting

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University Medical Center, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mikhail AI, Nagy PL, Manta K, Rouse N, Manta A, Ng SY, Nagy MF, Smith P, Lu JQ, Nederveen JP, Ljubicic V, Tarnopolsky MA. Aerobic exercise elicits clinical adaptations in myotonic dystrophy type 1 patients independently of pathophysiological changes. J Clin Invest. 2022 May 16;132(10):e156125. doi: 10.1172/JCI156125. PMID 35316212